CLINICAL TRIAL: NCT00377234
Title: Randomized, Open-label, Multi-center Study to Investigate Patient Preference on Dosing in Women With Postmenopausal Osteoporosis Treated With Once Monthly Ibandronate and Once Weekly Risedronate. A Six Month, Two-sequence and Two-period Crossover Study.
Brief Title: A Study Comparing Monthly Boniva (Ibandronate) and Weekly Risedronate in Women With Post-Menopausal Osteoporosis.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MA19547
Record Dates: First submitted 2006-09-15; First posted 2006-09-18 (Estimated); Results first posted 2015-07-22 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Post Menopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Risedronic Acid; Ibandronic Acid

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: ibandronate [Bonviva/Boniva]
- 2 (Active Comparator)
  Interventions: Drug: Risedronate

INTERVENTIONS:
Drug: Risedronate — 35mg po weekly for 12 weeks
  Arms: 2
Drug: ibandronate [Bonviva/Boniva] — 150mg po monthly for 3 months
  Arms: 1

SUMMARY:
This 2 arm crossover study will evaluate patient reported preference for either once monthly Boniva (150mg p.o.) or once weekly risedronate (35mg p.o.). Patients with post-menopausal osteoporosis will be randomized to receive Boniva for 3 calendar months or risedronate for 12 weeks; they will then cross over to receive the alternative treatment for a further 12 weeks/3 months. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* ambulatory women with post-menopausal osteoporosis;
* patients who are bisphosphonate-naive, or who have previously received oral daily or i.v. bisphosphonate therapy (fulfilling certain criteria detailed in the protocol).

Exclusion Criteria:

* malignant disease diagnosed within previous 10 years (except for successfully resected basal cell cancer;) breast cancer within previous 20 years;
* inability to stand or sit upright for at least 60 minutes;
* disease/disorder/treatment with drugs known to influence bone metabolism.

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2006-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (45):
- United States (45):
  - Birmingham, Alabama
  - Mesa, Arizona
  - Scottsdale, Arizona
  - Jonesboro, Arkansas
  - Anaheim, California
  - San Diego, California
  - Waterbury, Connecticut
  - Boynton Beach, Florida
  - Jupiter, Florida
  - Largo, Florida
  - Leesburg, Florida
  - Merritt Island, Florida
  - Ocala, Florida
  - Pembroke Pines, Florida
  - Spring Hill, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Douglasville, Georgia
  - Gainesville, Georgia
  - Marietta, Georgia
  - Madisonville, Kentucky
  - Bethesda, Maryland
  - Missoula, Montana
  - Omaha, Nebraska
  - Morehead City, North Carolina
  - New Bern, North Carolina
  - Jamestown, North Dakota
  - Cincinnati, Ohio
  - Mogadore, Ohio
  - Tulsa, Oklahoma
  - Duncansville, Pennsylvania
  - Erie, Pennsylvania
  - Feasterville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Anderson, South Carolina
  - Memphis, Tennessee
  - Selmer, Tennessee
  - Bedford, Texas
  - Bryan, Texas
  - Dallas, Texas
  - Houston, Texas
  - Temple, Texas
  - Richmond, Virginia
  - Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 488 patients who were screened, 356 patients were enrolled into the study at 44 centers in the USA and randomized to treatment with ibandronate and risedronate. One hundred eighty patients were randomized to Sequence A (Period 1 ibandronate, Period 2 risedronate), and 176 patients to Sequence B (Period 1 risedronate, Period 2 ibandronate).
Groups:
- Sequence A: Ibandronate followed by risedronate
- Sequence B: Risedronate followed by ibandronate
Period: Overall Study
Arm/Group | Sequence A | Sequence B
Started | 180 | 176
Randomized | 180 | 176
Did Not Receive Study Treatment | 3 | 2
Received Treatment | 177 | 174
Safety Analysis Set: Period 1 | 177 | 174
Safety Analysis Set: Period 2 | 153 | 150
Safety Analysis Set: Ibandronate | 177 | 150
Safety Analysis Set: Risedronate | 153 | 174
Completed | 146 | 145
Not Completed | 34 | 31
Not completed — Adverse Event | 14 | 17
Not completed — Withdrawal by Subject | 11 | 9
Not completed — Lost to Follow-up | 4 | 2
Not completed — Administrative | 2 | 1
Not completed — Not assigned | 3 | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence A | Sequence B | Total
Number analyzed (Participants) | 177 | 174 | 351
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.6 (7.0) | 64.0 (6.7) | 64.3 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 177 | 174 | 351
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 177 | 174 | 351

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Preferred Ibandronate Monthly Dosing to Risedronate Weekly Dosing
Description: Patients who had taken at least one dose of each study medication were asked to answer a Preference Questionnaire (answered by patients before any study procedures took place at the 6 month visit or at the early termination visit). The questionnaire included three questions on the preferred dosing schedule, and one question asking which schedule was more convenient. No assistance was allowed in completing the questionnaire.
Time Frame: at 6 months
Population: Modified Intent to Treat (mITT), defined as the safety analysis set excluding those participants who did not express a preference for one treatment
Measure: Number; unit: percentage of participants
Groups:
- During Sequence A: Ibandronate followed by risedronate
- During Sequence B: Risendronate followed by ibandronate
- Total: During period 1 + during period 2
Arm/Group | During Sequence A | During Sequence B | Total
Number analyzed (Participants) | 131 | 147 | 278
percentage of participants | 81.7 | 78.2 | 79.9
Statistical Analysis 1: Comparison: Total; Test type: Superiority or Other; p < 0.0001, Garts Test — Null hypothesis: Preference rate (including patients not expressing treatment preference and considering order treatments were received) for monthly ibandronate = 50%. Null hypothesis is rejected if P-value was below significance threshold of P <0.05
Statistical Analysis 2: Comparison: Total; Test type: Superiority or Other; p < 0.0001, Prescott Test — The reported p-values for the primary analysis test whether the overall preference rate for ibandronate equals 50%. Preference within each sequence is not tested

2. Secondary Outcome: Percentage of Participants Who Found Once-monthly Ibandronate to be More Convenient Than Once-weekly Risedronate
Description: as for outcome 1
Time Frame: within 6 months
Population: mITT, defined as the safety analysis set excluding those participants who did not express a preference for one treatment
Measure: Number; unit: percentage of participants
Groups:
- During Sequence B: Risedronate followed by ibandronate
Arm/Group | During Sequence A | During Sequence B | Total
Number analyzed (Participants) | 131 | 131 | 262
percentage of participants | 85.5 | 87.0 | 86.3

3. Secondary Outcome: Intensity of Upper Gastrointestinal (GI) Symptoms
Description: Patients were given a diary in which to record their upper GI events during the first 12 weeks of treatment. The diary was to be completed weekly and the occurrence of symptoms and their intensity recorded using a pre-defined list.
Time Frame: within 3 months
Population: Safety analysis set
Measure: Number; unit: percentage of participants
Groups:
- Ibandronate: While being treated with ibandronate
- Risedronate: While being treated with risendronate
Arm/Group | Ibandronate | Risedronate
Number analyzed (Participants) | 177 | 174
percentage of participants
  Any | 46.1 | 56.5
  Mild | 41.3 | 49.1
  Moderate | 32.3 | 36.0
  Severe | 15.6 | 12.4

4. Secondary Outcome: Mean Change From Baseline in Bone Resorption and Bone Formation Markers, Serum C-telopeptide of α-chain of Type I Collagen (CTX) and Bone Specific Alkaline Phosphatase (BSAP)
Description: During the conduct of this study, it came to the attention of the sponsor that mislabeling of blood samples for the analysis of the bone turnover markers, serum CTX and BSAP, had occurred at more than half of the 44 clinical trial sites. As a result of this mislabeling, the bone turnover marker samples could not be assigned correctly to the two time points at which they were collected (samples collected at baseline and those collected at the crossover visit which occurred after 3 months following the start of trial treatment). Thus, the results of bone turnover markers could not be reliably assessed. Therefore, summary tables showing the mean and median change from baseline for both serum CTX and BSAP for patients randomized to Sequence A (3 months of ibandronate followed by 12 weeks of risedronate) or Sequence B (12 weeks of risedronate followed by 3 months of ibandronate) are not presented, as a valid interpretation of the data cannot be made.
Time Frame: 3 months
Population: Mislabeling of blood samples for analysis of bone turnover markers resulted in inability to correctly assign samples to two time points at which they were collected (baseline and crossover visit). Results could not be reliably assessed or reported.
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Median Change From Baseline in Bone Resorption and Bone Formation Markers, Serum C-telopeptide of α-chain of Type I Collagen (CTX) and Bone Specific Alkaline Phosphatase (BSAP)
Description: as for outcome 4
Time Frame: 3 months
Population: as for outcome 4
Arm/Group | Sequence A | Sequence B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Study duration was approximately 6 months (3 months and 12 weeks) and a follow-up period of 15 days after the completion of treatment was included to assess safety information. Participants were assessed for adverse events for a total of 6.5 months.
Description: The safety analysis set is a modified intent to treat population, defined as all subjects who received the respective treatment.
Groups:
- Ibandronate: Ibandronate adverse events
- Risedronate: Risendronate adverse events
Arm/Group | Ibandronate | Risedronate
Serious Adverse Events (participants affected / at risk) | 5/327 | 3/327
Other Adverse Events (participants affected / at risk) | 0/327 | 0/327
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibandronate (N=327) | Risedronate (N=327)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Vitreous Haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Abdominal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ovarian Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Malignant Hypertension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.